CLINICAL TRIAL: NCT00744549
Title: The Impact of Antioxidants on MRI Markers of Cell Proliferation and Hypoxia Among Men on Active Surveillance With Early Stage Prostate Cancer
Brief Title: Study of Antioxidants on MRI Detectable Early Stage Prostate Cancer Among Men on Active Surveillance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Prostate Cancer Research Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0580-B
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Cancer of the Prostate; Prostate Cancer; Prostatic Neoplasms
Keywords: Male Urogenital Diseases; Antioxidants; Vitamin E; Vitamin D; Lycopene; Selenium
MeSH Terms: conditions — Prostatic Neoplasms; Male Urogenital Diseases | interventions — Lycopene; Cholecalciferol; Selenium; Tea; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): This group of men will be on active treatment (antioxidants) for one year and placebo for the second year.
  Interventions: Dietary Supplement: Lycopene, Vitamin D3, Selenium, Green Tea Extract, Vitamin E; Drug: Placebo
- B (Experimental): This group of men will be on placebo for one year and active treatment (antioxidants) for the second year.
  Interventions: Dietary Supplement: Lycopene, Vitamin D3, Selenium, Green Tea Extract, Vitamin E; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Lycopene, Vitamin D3, Selenium, Green Tea Extract, Vitamin E — Twice a day with meals. Lycopene - 20 mg, Vitamin D3 - 200 IU, Selenium - 100 mcg, Green Tea Extract - 75 mg, Vitamin E - 50 IU
Drug: Placebo — Twice a day with meals.

SUMMARY:
The purpose of this study is to determine whether antioxidants (vitamin E, selenium and lycopene)can change(reduce)prostate tumor size or blood flow to the prostate as determined by MRI imaging among men on Active Surveillance.

ELIGIBILITY:
Inclusion Criteria:

* MRI detectable prostate cancer
* PSA less than 15 ng/ml
* Gleason score <= 7
* Prostate cancer staging T1c or T2a

Exclusion Criteria:

* Concurrent use of high-dose vitamins which include selenium, lycopene, vitamin D or vitamin E
* Other malignancies diagnosed or requiring treatment within the past 5 years (except superficial bladder cancer or basal cell carcinoma)
* Current use of Proscar or Avodart

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the impact of combination vitamin E, lycopene, and selenium on MRI detected prostate tumor size and/or tumor blood flow among me on active surveillance | At baseline MRI compared to 1-year MRI compared to 2-year MRI

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network - Princess Margaret Hospital, Toronto, Ontario, Canada